CLINICAL TRIAL: NCT06874114
Title: REal-world EvideNce Study describinG treAtment Intensification Patterns amonG Canadian patiEnts With mHSPC Using EHR Data From Community Urology Clinics
Brief Title: An Observational Study to Learn More About Treatment Patterns and Factors Determining the Choice of Treatment in Canadian Men With Metastatic Hormone Sensitive Prostate Cancer in Routine Medical Care
Acronym: RE-ENGAGE
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22917
Record Dates: First submitted 2025-02-21; First posted 2025-03-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort A: No Androgen Deprivation Therapy (ADT) nor Androgen Receptor Pathway Inhibitor (ARPi) treatment
- Cohort B: Androgen Deprivation Therapy (ADT) Monotherapy: Patients initiating or continuing ADT alone for up to 180 days after Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) diagnosis
- Cohort C: Androgen Deprivation Therapy (ADT)+Docetaxel: Patients initiating docetaxel within 180 days of start of ADT after Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) diagnosis
- Cohort D: Androgen Deprivation Therapy (ADT)+Androgen Receptor Pathway Inhibitor (ARPi): Patients initiating ARPi within 180 days of start of ADT after mHSPC diagnosis
- Cohort E: Androgen Deprivation Therapy (ADT)+Androgen Receptor Pathway Inhibitor (ARPi)+Docetaxel: Patients initiating ARPi and docetaxel within 180 days start of ADT after Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) diagnosis

SUMMARY:
This is an observational study in which only data are collected from adult Canadian men with metastatic hormone sensitive prostate cancer (mHSPC) are studied. Participants will not receive any advice on treatment or any changes to the healthcare.

Metastatic hormone sensitive prostate cancer is a cancer of the prostate gland, a male reproductive gland found below the bladder. Metastatic means that cancer has spread to other parts of the body. Hormone-sensitive means it can be treated with anti-hormonal therapy such as androgen deprivation therapy (ADT).

ADT lowers the level of testosterone and slows down the growth of cancer cells. However, in some cases, ADT alone is not sufficient and doctors recommend combining it with treatments like Androgen Receptor Pathway Inhibitors (ARPi) and/or docetaxel to stop the growth of cancer cells.

ARPi slow down the growth of the cancer cells by blocking a sex hormone called the androgens from attaching to the protein found in the cancer cells. ARPi includes medicines like apalutamide, darolutamide, and enzalutamide.

Docetaxel is a medicine used to treat different types of cancer and works by stopping the growth and spread of cancer cells. ADT, ARPi, and docetaxel are approved treatments for men with mHSPC in Canada.

The participants in this study are already receiving treatment for mHSPC as part of their routine medical care from their doctors.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥ 18 years diagnosed with mHSPC verified by radiographic evidence of metastasis with Conventional Imaging (CI) or Prostate Specific Membrane Antigen-Positron Emission Tomography (PSMA-PET), and histologically confirmed carcinoma
* At least 6 months follow-up post-diagnosis period, unless the patient died earlier

Exclusion Criteria:

* ADT use for >6 months or any use of ARPi (ADT use in the neoadjuvant or adjuvant setting where the patient has been off treatment for 12 months or more is allowed)
* This criterion is to ensure that we are capturing mHSPC patients and not Metastatic Castration-Resistant Prostate Cancer (mCRPC) patients who have progressed from earlier stages
* Evidence of inclusion in clinical trials during the study period

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will include patients from 8 community urology clinics across two Canadian provinces. According to the Canadian Urological Association (CUA), community urologists are defined as non-academic institutions with considerably less access to residents, allied professional support, new technology, research funding, and/or continuous peer-review. Their referral base is primarily family physicians, and their teaching responsibilities include primarily family physicians and nurses.
  The 8 community urology clinics will be selected purposefully based on the specific data needs to address the study objectives, taking into consideration factors such as clinic size, and where possible, uptake of treatment intensification to increase the generalizability of the findings.
  However, it is acknowledged that this is a convenience sample, and may not accurately represent the wider mHSPC Canadian population.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment intensification in patients with mHSPC | January 2018 until June 2026
  The primary outcome of interest is utilization of treatment intensification in patients with mHSPC, including: Frequencies and percentages of patients in each treatment cohort

SECONDARY OUTCOMES:
Demographics: age in years | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: date of diagnosis of prostate cancer | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: date of mHSPC diagnosis (as confirmed by radiographic evidence of metastasis with CI or PSMA-PET, and histologically confirmed carcinoma) | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: year of mHSPC diagnosis | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: Eastern Cooperative Oncology Group (ECOG) score | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: Gleason score | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: comorbidities (Charlson Comorbidity Index) | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: disease volume/risk at baseline | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Clinical characteristics: radiological evidence of metastases (number and site) at time of initial mHSPC diagnosis | January 2018 until June 2026
  Data utilized consists of secondary-use data: all data used was collected as part of routine clinical practice (patients' medical records) prior to study initiation
Physician characteristics: practice size | January 2018 until June 2026
  Physician characteristics that are related to treatment intensification. Data was extracted from the EHR where available, and via communication with the clinicians.
Physician characteristics: years in practice | January 2018 until June 2026
  Physician characteristics that are related to treatment intensification. Data was extracted from the EHR where available, and via communication with the clinicians
Physician characteristics: number of patients seen annually with prostate cancer | January 2018 until June 2026
  Physician characteristics that are related to treatment intensification. Data was extracted from the EHR where available, and via communication with the clinicians
Physician characteristics: treatment areas of expertise | January 2018 until June 2026
  Physician characteristics that are related to treatment intensification. Data was extracted from the EHR where available, and via communication with the clinicians.
Reasons for treatment discontinuation and/or changing treatment by treatment cohort | January 2018 until June 2026
  Reasons for treatment discontinuation and/or changing treatment by treatment cohort, including:
  * Frequency and percentages of patients discontinuing/changing treatment due to AEs (and treatment-relatedness, if possible)
  * Frequency and percentages of patients discontinuing/changing treatment due to progression to mCRPC
  * Frequency and percentages of patients discontinuing treatment due to death
  * Frequency and percentages of patients discontinuing/changing treatment due to any other reason
Time to treatment discontinuation (TTD) | January 2018 until June 2026
  TTD will be measured from start of study treatment (index date 2) until discontinuation of ADT in monotherapy regimens or discontinuation of ARPi in doublet or triplet regimens or discontinuation of docetaxel within < 6 cycles in the docetaxel regimens. Treatment discontinuation will be defined as the last date treatment is given
mCRPC real-world progression free survival (rwPFS) | January 2018 until June 2026
  rwPFS will be measured from mHSPC diagnosis (index date 1) until date of progression as documented in physician notes or rising PSA levels (using PCW3 definition) despite castrate testosterone levels, where available, or date of death
Referral patterns for intensification among patients with mHSPC | January 2018 until June 2026
  Determine if the study can identify a pattern in which mHSPC patients can be candidates for intensification therapy, based on the patient data.
Docetaxel dosage adjustments | January 2018 until June 2026

CONTACTS AND LOCATIONS:
Locations (1):
- Pentavere, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Related Info — http://clinicaltrials.bayer.com/study/22917